CLINICAL TRIAL: NCT01251471
Title: Neural, Genetic, and Peripheral Correlates of SSRI Pharmaco-Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Lukas Pezawas, Lukas Pezawas, MD, Medical University of Vienna, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OENB-13903
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Depression
Keywords: major depressive disorder; MDD; imaging genetics; pharmacoMRI
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): Escitalopram, p.o., 10 mg/d; optional 20 mg/d after 2 weeks for 8 weeks
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10 mg/d; optional 20 mg/d after 2 weeks.
  Other Names: Lexapro; Cipralex; Seroplex; Lexamil

SUMMARY:
The aim of this pharmaco-MRI study is to investigate neural correlates of variable antidepressant treatment response driven by genetic variation in multiple genes involved in depression.

Thirty Major Depressive Disorder (MDD) patients with a concurrent major depressive episode will undergo three MRI scanning sessions after escitalopram treatment initiation. Furthermore, extensive behavioral assessments and measures of potential peripheral markers such lymphocyte mRNA or pharmacological parameters on platelets or lymphocytes will be performed.

Imaging measures have been suggested to be superior for drug response assessment as compared to psychometric scales, which hardly correlate with biological parameters. Since imaging techniques are too expensive and sophisticated for a broad clinical use, this study will provide pilot data on potential peripheral biomarkers of neural activation being related to drug response.

DETAILED DESCRIPTION:
The aim of this pharmaco-MRI study is to investigate neural correlates of variable antidepressant treatment response driven by genetic variation in multiple genes involved in depression.

Thirty Major Depressive Disorder (MDD) patients with a concurrent major depressive episode will undergo three MRI scanning sessions at baseline, 4 hours and 8 weeks after escitalopram treatment initiation. During each MRI session, one structural and 3 fMRI scans each engaging different brain circuitries will be performed. All subjects will undergo extensive behavioral assessment and will be genotyped. Furthermore, potential peripheral markers such lymphocyte mRNA or pharmacological parameters on platelets or lymphocytes will be assessed.

The investigators expect that genetic variants which have been associated with variable response to SSRIs in previous Imaging Genetics studies are modulating neural targets of drug response. Moreover, peripheral markers are expected to correlate with these brain region measurements.

Imaging measures have been suggested to be superior for drug response assessment as compared to psychometric scales, which hardly correlate with biological parameters. Since imaging techniques are too expensive and sophisticated for a broad clinical use, this study will provide pilot data on peripheral biomarkers of neural activation being related to drug response. Furthermore, this study will demonstrate whether and how genotypes impact on the dynamics of neural drug response in vivo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 -45 years
* Right-handedness
* DSM-IV diagnosis of a major depressive episode (SCID)
* a MADRS score ≥20 and ≤ 30
* ability to be managed as outpatients
* ability to fulfill the criteria to undergo an MRI scan
* Caucasian subjects of European ancestry

Exclusion Criteria:

* previous or concurrent major medical or neurological illness
* clinically significant abnormal values in routine laboratory screening or general physical examination
* DSM-IV diagnosis of substance dependence within the past year, except for caffeine or nicotine or current substance abuse
* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or an anxiety disorder as a primary diagnosis
* the use of any psychotropic drug within the last two months unresponsiveness of a former major depressive episode to an adequate antidepressive drug dosing of at least 6 weeks duration or any kind of therapy resistance
* a history of severe drug allergy or hypersensitivity or known hypersensitivity to escitalopram
* being acutely suicidal either indicated by a score ≥ 5 on item 10 (suicidal thoughts) on the MADRS or a score ≥ 4 on the HAM-D 21 (suicidal thoughts) or according to the investigator´s opinion
* failures to comply with the study protocol or to follow the instructions of the investigating team
* current pregnancy or breast feeding
* metallic implants or other contraindications to MRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
BOLD signal | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Pezawas, MD, Principal Investigator — Medical University of Vienna, Dept. of Psychiatry and Psychotherapy
Locations (1):
- Medical University of Vienna, Dept. of Psychiatry and Psychotherapy, Vienna, Vienna, Austria

REFERENCES:
- [Background] Scharinger C, Rabl U, Sitte HH, Pezawas L. Imaging genetics of mood disorders. Neuroimage. 2010 Nov 15;53(3):810-21. doi: 10.1016/j.neuroimage.2010.02.019. Epub 2010 Feb 13. PMID 20156570
- [Background] Pezawas L, Meyer-Lindenberg A. Imaging genetics: Progressing by leaps and bounds. Neuroimage. 2010 Nov 15;53(3):801-3. doi: 10.1016/j.neuroimage.2010.08.001. No abstract available. PMID 20816317
- [Background] Rabl U, Scharinger C, Muller M, Pezawas L. Imaging genetics: implications for research on variable antidepressant drug response. Expert Rev Clin Pharmacol. 2010 Jul;3(4):471-89. doi: 10.1586/ecp.10.35. PMID 22111678
- See also: Dep. Psychiatry and Psychotherapy — http://www.meduniwien.ac.at/psychiatrie/